CLINICAL TRIAL: NCT04465006
Title: Efficacy of Hippotherapy Simulator Exercise Program in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2018.425
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Hippotherapy; Cerebrovasculer disorders; Stroke Rehabilitation; Balance; Exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group received hippotherapy exercise, while the other group received conventional exercise.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hippotherapy Simulator Group (Experimental): Getting a diagnosis of stroke by a specialist physician, Being between the ages of 18-65, Having a stroke history of 3- 36 months, To be able to sit without support while both soles are in contact with the floor, To be able to walk independently with or without using walking aid, To be able to understand and follow audio and visual warnings, Scoring 24 points or more from the Mini Mental State Exam.
  Interventions: Other: Hippotherapy Simulator
- Conventional Exercise Group (Experimental): Getting a diagnosis of stroke by a specialist physician, Being between the ages of 18-65, Having a stroke history of 3- 36 months, To be able to sit without support while both soles are in contact with the floor, To be able to walk independently with or without using walking aid, To be able to understand and follow audio and visual warnings, Scoring 24 points or more from the Mini Mental State Exam.
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Hippotherapy Simulator — Patients in the hippotherapy simulator group received 30 sessions of treatment for 6 weeks, 5 days a week and 1 hour a day. 45 minutes of Neurodevelopmental treatment exercises and 15 minutes of hippotherapy simulation exercise program were applied to the participants in this group.
  Arms: Hippotherapy Simulator Group
Other: Conventional Exercise — Patients in the conventionnal exercise group received 30 sessions of treatment for 6 weeks, 5 days a week and 1 hour a day. 60 minutes of Neurodevelopmental treatment exercises were applied to the participants in this group.
  Arms: Conventional Exercise Group

SUMMARY:
The aim of our study is to investigate the effects of hippotherapy simulator exercises in addition to the conventional rehabilitation program on the balance, postural control, mobility, functional capacity, and independence levels of stroke patients.

DETAILED DESCRIPTION:
Twenty-six 18- 65 years of patients with stroke were included in the study. Patients were divided into two groups as hippotherapy simulator group (HSG) (n = 13) and conventional exercise group (CEG) (n = 13). Patients were evaluated with Berg Balance Scale (BBS) for balance, Postural Assessment Scale for Stroke (PASS) for postural control, Rivermead Mobility Index (RMI), and Time Up- Go Test (TUG) for mobility, 2min. Walking Test (2mWT) for functional capacity and Barthel Index (BI) for the level of independence respectively before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Getting a diagnosis of stroke by a specialist physician,
* Being between the ages of 18-65,
* Having a stroke history of 3- 36 months,
* To be able to sit without support while both soles are in contact with the floor,
* To be able to walk independently with or without using a walking aid,
* To be able to understand and follow audio and visual warnings,
* Scoring 24 points or more from the Mini-Mental State Exam.

Exclusion Criteria:

* Multiple stroke stories,
* Hemorrhagic type stroke history,
* Those with a history of falling in the past 1 year,
* Those with a history of epilepsy,
* Uncontrolled history of Hypertension and Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Day 0 - Day 45
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Postural Assessment Scale for Stroke | Day 0 - Day 45
  It measures the ability of an individual with stroke to maintain stable postures and equilibrium during positional changes. It consists of a 4-point scale where the items are scored from 0 to 3, and the total scoring ranges from 0 to 36
Rivermead Mobility Index | Day 0 - Day 45
  The Rivermead Mobility Index assesses functional mobility in gait, balance and transfers after stroke.
Timed Up and Go Test | Day 0 - Day 45
  The Timed Up and Go (TUG) test is a performance-based measure of functional mobility that was initially developed to identify mobility and balance impairments in older adults.
2 Minute Walk Test | Day 0 - Day 45
  2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity.
Barthel Index | Day 0 - Day 45
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL).

CONTACTS AND LOCATIONS:
Overall Officials: Zubeyir Sarı, Assoc Prof, Study Chair — Department of Physiotherapy and Rehabilitation - Marmara University; Sergen Ozturk, PT, Principal Investigator — Department of Physiotherapy and Rehabilitation - Marmara University
Locations (1):
- Private Ersoy Hospital, Sultanbeyli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson W, Onuma O, Owolabi M, Sachdev S. Stroke: a global response is needed. Bull World Health Organ. 2016 Sep 1;94(9):634-634A. doi: 10.2471/BLT.16.181636. No abstract available. PMID 27708464
- [Background] Nedeltchev K, der Maur TA, Georgiadis D, Arnold M, Caso V, Mattle HP, Schroth G, Remonda L, Sturzenegger M, Fischer U, Baumgartner RW. Ischaemic stroke in young adults: predictors of outcome and recurrence. J Neurol Neurosurg Psychiatry. 2005 Feb;76(2):191-5. doi: 10.1136/jnnp.2004.040543. PMID 15654030
- [Background] Huang CY, Lin GH, Huang YJ, Song CY, Lee YC, How MJ, Chen YM, Hsueh IP, Chen MH, Hsieh CL. Improving the utility of the Brunnstrom recovery stages in patients with stroke: Validation and quantification. Medicine (Baltimore). 2016 Aug;95(31):e4508. doi: 10.1097/MD.0000000000004508. PMID 27495103
- [Result] Kim S, Yuk GC, Gak H. Effects of the horse riding simulator and ball exercises on balance of the elderly. J Phys Ther Sci. 2013 Nov;25(11):1425-8. doi: 10.1589/jpts.25.1425. Epub 2013 Dec 11. PMID 24396203
- [Result] Ciou SH, Hwang YS, Chen CC, Chen SC, Chou SW, Chen YL. Balance training using an interactive game to enhance the use of the affected side after stroke. J Phys Ther Sci. 2015 Dec;27(12):3855-61. doi: 10.1589/jpts.27.3855. Epub 2015 Dec 28. PMID 26834368